CLINICAL TRIAL: NCT06701487
Title: SFB TRR 265: Losing and Regaining Control Over Drug Intake Work Package 1 of Project B03: General and Specific Pavlovian-to-Instrumental Transfer Effects in a Range of Substance Use Disorders
Brief Title: Role of Pavlovian Mechanisms for Control Over Substance Use
Acronym: ReCoDe
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Charite University, Berlin, Germany (Other); Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Other Study IDs: 40217046121
Record Dates: First submitted 2024-09-25; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Use Disorder (AUD); Alcoholism; Substance Use Disorders; Cannabis Use Disorder; Methamphetamine-dependence; Amphetamine Use Disorder; Cocaine Use Disorder
Keywords: Substance Use Disorder (SUD); Cannabise Use Disorder; Methamphetamine Use Disorder; Amphetamine Use Disorder; Cocaine Use Disorder; Alcohol Use Disorder (AUD); Pavlovian-to-Instrumental Transfer (PIT); General Pavlovian-to-Instrumental Transfer; Outcome-specific Pavlovian-to-Instrumental Transfer; Amygdala; Ventral Striatum; Neuroimaging; Humans; Surveys and Questionnaires; Reward; Cues
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Alcohol use disorder (AUD): Participants with alcohol use disorder (moderate to severe if no withdrawal symptoms) and no other substance use disorder (SUD)
  Interventions: Biological: fMRI imaging (BOLD); Biological: sMRI (structure); Behavioral: Pavlovian-to-instrumental transfer (PIT) paradigm; Diagnostic Test: Basic psychological assessment (interview); Diagnostic Test: Basic psychological assessment (questionnaires); Behavioral: Neuropsychological tests
- Alcohol use disorder (AUD) and Substance use disorder (SUD): Participants with Alcohol use disorder (AUD) and comorbid Substance use disorder (SUD) (moderate to severe cases without withdrawal symptoms) including:
  Participants with alcohol use disorder (AUD) and/or cannabis use disorder and/or methamphetamine use disorder and/or amphetamine use disorder and/or cocaine use disorder.
  Interventions: Biological: fMRI imaging (BOLD); Biological: sMRI (structure); Behavioral: Pavlovian-to-instrumental transfer (PIT) paradigm; Diagnostic Test: Basic psychological assessment (interview); Diagnostic Test: Basic psychological assessment (questionnaires); Behavioral: Neuropsychological tests
- Non-AUD Substance use disorder (SUD): Participants with substance use disorder (moderate to severe cases without withdrawal symptoms) without alcohol use disorder (AUD) including:
  Participants with methamphetamine use disorder and/or cannabis use disorder and/or amphetamine use disorder and/or cocaine use disorder
  Interventions: Biological: fMRI imaging (BOLD); Biological: sMRI (structure); Behavioral: Pavlovian-to-instrumental transfer (PIT) paradigm; Diagnostic Test: Basic psychological assessment (interview); Diagnostic Test: Basic psychological assessment (questionnaires); Behavioral: Neuropsychological tests
- Control group: Healthy participants without AUD or SUD
  Interventions: Biological: fMRI imaging (BOLD); Biological: sMRI (structure); Behavioral: Pavlovian-to-instrumental transfer (PIT) paradigm; Diagnostic Test: Basic psychological assessment (interview); Diagnostic Test: Basic psychological assessment (questionnaires); Behavioral: Neuropsychological tests

INTERVENTIONS:
Biological: fMRI imaging (BOLD) — Will be used to investigate neural correlates of Pavlovian-to-instrumental transfer (PIT) effects by measuring the blood oxygenation level dependent (BOLD) response of neural activation in the mesolimbic system.
Biological: sMRI (structure) — Will be used to investigate neural correlates of PIT effects by identifying abnormalities in cortical gray and white matter volume.
Behavioral: Pavlovian-to-instrumental transfer (PIT) paradigm — The paradigm consists of four parts:
  In the first part, an instrumental learning task is completed in which subjects must learn which stimuli require a response and which do not. In the second part, a classical (Pavlovian) conditioning task is then completed in which subjects learn by passive viewing which stimuli are associated with certain amounts of money. The third part measures to which instrumental responses (learned in Part 1) are modulated by the presentation of the classically conditioned stimuli (learned in Part 2). At the same time drug-associated stimuli are presented in the background measuring to which extent they conflict with the learned instrumental behavior. In the last part, query trials are implemented in which the participants have to choose between two pictures to assess the relative cue value.
Diagnostic Test: Basic psychological assessment (interview) — * Alcohol, Smoking and Substance Involvement Screening Test (ASSIST)
  * Quantity Frequency: Alcohol, Cannabis, (Meth-) Amphetamine, Cocaine)
  * SCID: AUD and SUD (Cannabis, Methamphetamine, Amphetamine, Cocaine) criteria and last year & depressive symptoms & symptoms for Mania and psychotic disorder (acute and lifetime) MiniDIPS psychotic disorders
Diagnostic Test: Basic psychological assessment (questionnaires) — * Sociodemographics
  * Edinburgh Handedness Inventory (EHI)
  * Fagerström Test for Nicotine depend (FTND)
  * Barratt Impulsiveness Scale - Kurzversion (BIS-15)
  * Allgemeine Depressionsskala (ADS)
  * State-Trait-Anxiety Inventory (STAI-T and STAI-S)
  * Adult ADHD Self-Report Scale (ASRS)
  * Alcohol Use Disorders Identification Test (AUDIT)
  * CAS -A (Alkohol)
  * Cannabis Use Disorders Identification Test (CUDIT)
  * Fragebogen zu Gedanken und Gefühle 14 Items (FGG-14)
  * Fragebogen zur Sozialen Unterstützung (F-SozU-K14)
  * Trierer Inventar zum chronischen Stress (TICS)
  * Oslo 3-Items-Social-Support Scale (Oslo-3)
  * Social Readjustment Rating Scale (SRRS)
  * International Trauma Questionnaire (ITQ)
  * Positive and Negative Affect Schedule (PANAS)
Behavioral: Neuropsychological tests — * Digit-Symbol-Test (DST)
  * Digit Span Task
  * Value-based decision-making task (VBDM)

SUMMARY:
During the first funding period (1st FP), the investigators developed a novel full Pavlovian-to-instrumental transfer (PIT) task that allows assessing both, general and specific PIT to investigate whether specific PIT differs between alcohol use disorder (AUD) and control subjects. Preliminary analyses of the full transfer task indicate that AUD participants exhibit a stronger specific PIT effect compared to controls. Based on these findings, the investigators want to compare specific and general PIT effects in patients with moderate to severe substance use disorders (alcohol, cannabis, methamphetamine, amphetamine and cocaine) to healthy controls on the behavioral and neural level (fMRI).

DETAILED DESCRIPTION:
This projects research aim:

1. The investigators aim to compare general and specific PIT effects in patients with moderate to severe substance use disorder (Alcohol, Methamphetamine, Amphetamine and Cocaine) and healthy controls using the newly developed (1st FP) full transfer task and fMRI The investigators expect enhanced general PIT effects in patients compared to controls at the behavioral level, and at the neuronal level enhanced PIT-associated activations in the striatum, and lower activation in the prefrontal cortex (e.g., dlPFC).

The investigators expect enhanced general PIT effects in patients with multiple SUD compared to patients with single SUD.

The investigators expect increased behavioral and neuronal alcohol-specific PIT effects in patients groups that also meet AUD criteria compared to controls and to patients without AUD.

The investigators expect stronger behavioral and neural PIT effects (both general and specific) to predict more substance use at 3-month follow-up.

Therefore, the investigators aim to conduct the Experiments with the following Hypotheses:

Here the investigators assess on a behavioral and neural level a general and specific PIT task by using the full transfer task which was developed in the 1st FP and allows the assessment of both PIT tasks in one paradigm. This task consists of 4 parts: instrumental training, Pavlovian conditioning, Pavlovian-to-instrumental transfer phase and query trials to test participants' explicit knowledge.

The investigators will investigate HCs and three patient groups of high clinical relevance: Patients with (1) AUD without comorbid SUD (cannabis, methamphetamine, amphetamine or cocaine), (2) AUD with comorbid SUD (cannabis and/or methamphetamine and/or amphetamine and/or cocaine), (3) SUD (cannabis and/or methamphetamine and/or amphetamine and/or cocaine) without AUD. The investigators will recruit patients through the addiction outpatient clinic of the Charité (mainly cannabis), the special outpatient clinic for MUD at the University Hospital Dresden as well as the investigators' strategic partner clinic in Radebeul und Städtisches Klinikum Dresden. Furthermore, the investigators will be recruiting from the general population using advertisement. On site, they undergo the comprehensive assessment implemented for the TRR cohort during the 1st FP. The full PIT paradigm is applied as described in Figure 3. Three months after the examination, an online follow-up on the clinical course will be done by using redcap-based questionnaires.

Methods:

WP1 will follow an ANOVA with four groups, including post-hoc group differences.

Functional imaging data will be conducted using a 3 T MR scanner to acquire gradient echo t2*-weighted echo-planar images (EPI) and analyzed with SPM12. EPI images will be preprocessed and analyzed as implemented during the 1st FP.

Expected results:

The investigators expect that general PIT effects are increased in all patient groups vs. HCs. Moreover, the investigators expect that patients with AUD + comorbid SUD have greater general PIT effects than patients with AUD alone. Concerning alcohol specific PIT, the investigators expect that both AUD groups, but not patients with SUD without AUD have greater effects than HCs. Moreover, the investigators expect that patients with AUD + comorbid SUD have greater alcohol specific PIT effects than patients with AUD alone. Concerning neuroimaging, the investigators expect greater activations in striatum and reduced activation in the DLPFC during PIT in all patient groups vs. HCs. Moreover, the investigators expect greater activations in striatum and reduced activation in the DLPFC in patients with AUD + comorbid SUD as well as in patients with AUD alone. Of note, the investigators expect similar neural activations during specific PIT in HCs and patients with SUD without AUD.

Hypothesis 1a.:

General PIT effects are increased in all patient groups vs. HCs. Specifically, patients with AUD + comorbid SUD will show greater general PIT effects than patients with AUD alone. At the neuronal level patients will show enhanced PIT-associated activations in the striatum, and lower activation in the prefrontal cortex (e.g., dlPFC).

Hypothesis 1b:

Concerning alcohol specific PIT, it is expected that both AUD groups, but not patients with SUD without AUD have greater effects than HC. Moreover, patients with AUD + comorbid SUD will have greater alcohol specific PIT effects than patients with AUD alone. Moreover, the investigators expect greater activations in striatum and reduced activation in the DLPFC in patients with AUD + comorbid SUD as well as in patients with AUD alone.

Hypothesis 1c:

The investigators expect that enhanced specific and general PIT effects are associated with increased substance use at the 3-month follow-up.

Alternative strategies: In case of doubt about the extent to which gustatory alcohol and juice rewards increase the PIT effect in subjects with comorbid SUD, the investigators might alternatively develop and pilot a specific PIT paradigm with substance-related pictures.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18-65 years of age,
* AUD, and/or SUD subjects only: meet 4 or more criteria for DSM-5 alcohol-related and/or substance-related (cannabis, amphetamine, methamphetamine or cocaine disorder (not requiring withdrawal as assessed by an independent psychiatrist),
* Currently using alcohol without a desire for abstinence
* Ability to consent to the study and complete the questionnaires.
* Sufficient language(German) and motor skills for using PC
* existing health insurance

Exclusion Criteria:

* Lifetime diagnosis of DSM-5 bipolar disorder or schizophrenia or schizophrenia spectrum disorder (if induced by drugs, it should happen more than a month ago)
* Current threshold DSM-5 diagnosis of major depressive disorder, or presence of suicidal intention
* High risk (≤ 26) ASSIST scores in other substances other than alcohol, amphetamine, methamphetamine, cannabis, cocaine, tobacco
* History of traumatic brain injury or severe neurological disease (such as Dementia, Parkinson's disease, multiple sclerosis, Epilepsy, Meningitis, Stroke)
* Pregnancy or breastfeeding,
* Ingestion of medications known to interact with the dopamine system in the 10-day period prior to study participation or less than 4 half-lives after last ingestion (rapid urine test); A detailed list of permitted medication can be added upon request
* MR contraindications (e.g., pacemakers, metallic or electronic implants, metallic splinters, surgical staples)
* Color vision deficiency
* sensorineural hearing loss of 30 dB or greater,
* Tinnitus and
* Acute alcohol, substance (cannabis, or methamphetamine, amphetamine, cocaine) intoxication at assessement day verified by breath alcohol tests and drug intoxication verified by rapid urine test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Groups will be recruited through the addiction in- and outpatient clinic of the Charité, and from the special outpatient clinic for MUD at the University Hospital Dresden as well as from our strategic partner clinic in Radebeul and Städtisches Klinikum Dresden. Moreover, collaborating clinics in Berlin and Dresden will be recruited (with in- or outpatient clinics for treating patients with substance use disorder). Finally, we recruit persons from information centers for substance related problems and addiction groups in Berlin and Dresden and from the general population using advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Neural PIT effect | 1 day
  Blood oxygenation level dependent (BOLD) response, investigation of neuronal activation of the mesolimbic system in AUD patients and controls using 3 Tesla magnetic resonance imaging
Behavioral full-lever specific and general PIT effect | 1 day
  Strength of specific and general PIT effect assessed with the full-lever PIT paradigm.
  Specific: average percentage of alcohol choice difference during the presentation of alcohol or non-alcohol Pavlovian background. General: differences in number of button presses during the presentation of positive (+10 Euro) and negative (-10 Euro) Pavlovian backgrounds.

SECONDARY OUTCOMES:
Alcohol and Substance (cannabis, stimulant/cocaine) consumption after 3 months | 3 months after testing for behavioral and neural PIT effects
  Alcohol drinking amount and substance (cannabis, amphetamine, cocaine) consuming amount (quantity, frequency) during a follow-up period of 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Technische Universität Dresden, Dresden, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Belanger MJ, Chen H, Hentschel A, Garbusow M, Ebrahimi C, Knorr FG, Zech HG, Pilhatsch M, Heinz A, Smolka MN. Development of Novel Tasks to Assess Outcome-Specific and General Pavlovian-to-Instrumental Transfer in Humans. Neuropsychobiology. 2022;81(5):370-386. doi: 10.1159/000526774. Epub 2022 Nov 14. PMID 36380640